CLINICAL TRIAL: NCT03152877
Title: Efficacy of Extended-Release Liposomal Bupivacaine for Post-Partum Pain Management Following Obstetrical Laceration: A Prospective, Randomized, Single-Blinded Trial
Brief Title: Efficacy of Extended-Release Liposomal Bupivacaine for Post-Partum Pain Management Following Obstetrical Laceration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Katherine Dengler, MD, FPMRS Fellow, WRNMMC, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 216440
Record Dates: First submitted 2017-05-10; First posted 2017-05-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Pain, Obstetric
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposomal bupivacaine treatment group (Experimental): 20cc of liposomal bupivacaine will be injected into the vaginal/perineal laceration site, in subjects in the experimental arm, following completion of the surgical repair.
  Interventions: Drug: Bupivacaine Liposome Injectable Product
- 0.25% plain bupivacaine treatment group (Active Comparator): 20cc of 0.25% plain bupivacaine will be injected into the vaginal/perineal laceration site, in subjects in the active comparator arm, following completion of the surgical repair.
  Interventions: Drug: 0.25% plain bupivacaine

INTERVENTIONS:
Drug: Bupivacaine Liposome Injectable Product — 20cc of liposomal bupivacaine will be injected into the vaginal/perineal laceration site, once, following completion of the surgical repair.
  Other Names: Exparel
  Arms: Liposomal bupivacaine treatment group
Drug: 0.25% plain bupivacaine — 20cc of 0.25% plain bupivacaine will be injected into the vaginal/perineal laceration site, once, following completion of the surgical repair.
  Arms: 0.25% plain bupivacaine treatment group

SUMMARY:
We propose a prospective, randomized, single blinded trial with subjects recruited from the WRNMMC Labor and Delivery Unit to study post-partum efficacy of Exparel® for pain control in patients undergoing a vaginal delivery who sustained a second, third, or fourth degree obstetrical laceration. Subjects who meet inclusion criteria and agree to participate in the study will be consented upon admission for active labor or induction of labor and will be randomized to receive either 20mL of liposomal bupivacaine or 20ml of 0.25% plain bupivacaine, infiltrated through the perineum at completion of their obstetrical repair. Current standard of care is to receive no injection of local anesthetic upon completion of the repair.

The primary aim of the trial will be to evaluate post-partum pain using a visual analogue pain scale at days 1, 3 and 7 postpartum. All subjects will have acetaminophen, a non-steroidal anti-inflammatory drug and narcotic pain medication available for pain control regardless of assignment, which is the usual post-partum pain control regimen.

We anticipate a 30% difference in post-operative pain measurements between the Exparel® group and the plain bupivacaine group. Other aims of this study are to evaluate total medication usage, comparing the study group to the control, and compare quality of life measures between the two study groups.

DETAILED DESCRIPTION:
All pregnant female subjects over the age of 18 eligible to deliver vaginally at WRNMMC will be screened for potential recruitment in our long-acting liposomal bupivacaine (Exparel®) postpartum pain medicine trial prior to admission for active labor or induction of labor. At the 36 or 38 week visit, all pregnant patients will receive an information sheet describing the study participation and they will be asked to consider participating in the study. At the time of admission, patients will be asked if they were provided the study information sheet and if they would like to consent to study participation. Discussion of the study will occur after the delivery consent form for obstetric services has been signed and when discussion of postpartum pain management is addressed. Those subjects who meet inclusion criteria for the study will be randomized to either the plain bupivacaine group or exparel group after vaginal delivery and identification of a second, third, or fourth degree laceration.

Potential study subjects will be informed that the purpose of the study is to evaluate the efficacy of two different formulations of bupivacaine, 0.25% plain bupivacaine and liposomal bupivacaine (Exparel®) on postpartum pain following repair of a second, third, or fourth degree laceration sustained during vaginal delivery. This medication is FDA (Food and Drug Administration) approved and is currently being used in our hospital by other surgical sub-specialties as part of a multi-modal approach to post-operative pain control.

If a potential subject chooses to participate, she will be randomized to one of two groups, either a 0.25% bupivacaine injection of total 20 ml or an injection of total 20 ml long-active liposomal bupivacaine that will be injected in the subject's perineum (the tissue between the opening of the anus and the vagina) at the completion of the case in the delivery room. Regardless of the decision to participate in the study or which treatment group assignment, all subjects will have the same options for partum pain medications. There is no monetary payment for joining the study and subjects may choose to leave the study at any point during the study without consequence. They will still receive the same high standard of care from our Service.

The study is designed as a single blind, randomized study. This means the subject will not know which group a subject is assigned to until completion of the study. Subjects may choose to have their allocated study arm disclosed at this time. Randomization will occur using a computer-generated randomization program carried out in the Investigational Pharmacy by Dr. Moussavian. Subjects will be randomly assigned to either receive the study medication or bupivacaine.

The primary goal of the study is to assess how effective the study medication is in providing adequate pain control following repair of a second, third, or fourth degree laceration; therefore, the subjects' post-partum pain will be assessed at various intervals following the repair. On post-partum day one, subjects will be asked questions regarding their pain level in the vaginal area according to an 11-point visual pain scale. Subjects will also be asked about their bowel movements and any associated pain, again, using the same visual pain scale. Subjects will also be asked to the impact the pain has on 4 quality of life measures using an 11-point visual pain scale. Subjects will also be called or contacted via email thru Relay Health on post-op day three and on post-op day seven to assess pain on those days. Part of the study's goal is to assess whether the study medication provides pain control for longer than the acute (24 hour) period. Subjects will be given a visual pain scale to go home with so that they can reference it during their post-operative phone or email follow ups. Additionally, subjects will be asked to gather their pain medication bottles in order to count out the remaining pills in each bottle. This will allow us to determine the amount of oral pain medication used since discharge from the hospital.

Study participants will review the study consent form in detail with a provider, also an Associate Investigator in the study. The subject will be given a copy of the signed consent and a copy will remain on file in the patient's hospital record. The data sheet with non-identifiable subject number will be the only identifying information on the sheet. The subject's demographic data (gravida/parity, age, BMI, past medical history, allergies, current medications, history of significant drug or alcohol dependence) will be annotated on this data sheet along with the postpartum pain medications she receives. The data sheets will be kept in a locked cabinet within the resident library on the Labor and Delivery Unit, in a room locked during all-hours. A master list of subjects' full names and sponsor's last four of the social security number will be kept in the same location to reference the subjects' identification code. The dates of enrollment will be annotated on the master list as well. Follow-up phone call dates/email replies will be collected as well. Subjects will be re-assured that her participation in the study will be completely confidential and her identifying information will be double-locked when not being reviewed.

Following review of the study and obtaining of a consent form, the pain scale on the visual analog pain scale will be reviewed with the subject. Subjects must be willing to speak with a member of the study team on post-delivery day one, three, and seven regarding their post-operative pain, medications and bowel movements. Completion of day one data will occur in the hospital, prior to hospital discharge. The subject will be asked to indicate whether they prefer contact via phone or by email, using the Relay Health Network for day three and seven. A maximum of three attempts will be made to contact the subject on their designated follow up date, between the hours of 0800 and 2000. At the conclusion of the admission process, the subject will be reassured that if they desire removal from the study at any time, there will be no change in their customary post-delivery care.

At completion of the repair of the vaginal laceration, the consenting physician will enter the appropriate information on the data sheet, including the prescribed medications and quantities. A randomization envelope will be opened, assigning the patient to either the bupivacaine group or the Exparel group. The appropriate study medication will be obtained from the study refrigerator in the resident library and brought to the delivery room. Dr. Moussavian will randomize each subject to either Exparel or bupivacaine group, via pre-sealed opaque envelopes, and blind three 10mL syringes containing a total of 20 mL of either normal saline or liposomal bupivacaine (increments of 9mL, 9mL and 2mL). Syringe barrels will be covered with solid white labels to mask syringe contents. She will also print out a label to accompany the syringe to the Operating Room on the day of surgery stating:

"This subject is enrolled in study protocol #_______ and is to receive no additional bupivacaine post-operatively for 96 hours. "

This label will be placed on a wristband, following randomization, and will be worn during the entire hospital stay. It will assure that those subjects who receive liposomal bupivacaine will not receive additional bupivacaine but will still maintain blinding of all involved in the protocol.

On the day of admission for delivery, a member of the research team will, consent interested subjects for study participation. Any last minute questions can be answered and the subject will be advised that they can withdraw from the study at any time.

In the delivery room, the delivery team will identify the laceration and perform a repair, using standard technique. The use of 1% lidocaine with epinephrine may be used as a distention media to assist with pain relief during the repair so long as a minimum of 20 minutes elapses prior to injection of the study medication or bupivacaine. Once a laceration has been identified, a research team member will leave the room and obtain a randomization envelope from the locked study medication refrigerator in the residents' office. The envelope will be opened; identifying which treatment arm the patient will be assigned. The team member will come back to the room and tell the delivery nurse to leave the room and draw up the study medication into 20ml blinded-syringe. Once all surgical procedures have been completed, the circulating room nurse will verify the subject's name and date of birth and hand the 20mL blinded syringe to the delivering provider, who will attach an injection needle to the syringe. The surgeon will identify the bilateral perineal areas to be injected, approximated 1-2 cm below the opening of the vagina and 1-2 cm on either side of midline. 9 mL of the syringe solution will be injected into each bilateral location and then 2 mL at edge of vaginal opening (see figure1 below). The injection of the solution will occur at the completion of the surgical case. Following administration of the injection, the team will resume normal post-procedure care. The operating surgeon will verify the study protocol identification sticker has been placed in the subject's paper chart.

Post-delivery, the subject will recover in the delivery room per WRNMMC protocol and be transferred to either the postpartum unit as per routine post-operative criteria. Postpartum pain control will be managed by the obstetric team. Further injections of pain medications will not be given in the perineal area outside of the operating room.

On postpartum day one, a member of the obstetric team will visit the subject in order to obtain a pain and quality of life rating (0-10) based on the visual analog pain and quality of life scales. This will be documented as Day one data. Upon discharge postpartum care instructions will be reviewed and the subject will be reminded to expect her follow-up phone call or email via Relay Health on day three and seven.

During postpartum follow up on day 3 and day 7, subjects will be asked to get out their visual analog pain scale and rate the pain on their abdomen and the pain in the vagina on a 0-10 scale. The subject will also be asked if they have had a bowel movement and whether or not it was painful, based on the same pain scale 0-10. Subjects will be sent home with a copy of the pain scale with the hospital post-operative discharge paperwork. At postpartum phone or email contacts, subjects will be asked to count their remaining pain pills and these numbers will be documented in the data collection sheet.

All data sheets will be collected at the completion of each postpartum day and placed in the locked cabinet. Obstetric team members will have access to sheets to record data as it is collected. The data sheets will be shredded and disposed in a HIPAA compliant receptacle per WRNMMC protocol at the completion of the study. All consents and HIPAA authorizations will be maintained for six years after the study is closed. The Principal Investigator, Dr. Christopher Strauchon, will be available for debriefing of any subject after the study is completed if the subject desires.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females >18 years of age who sustained a second, third, or fourth degree laceration during a vaginal delivery, or operative vaginal delivery (forceps-assisted or vacuum-assisted) at Walter Reed National Military Medical Center

Exclusion Criteria:

* Known allergy to amide local anesthetics
* Unstable cardiac arrhythmia
* Hepatic impairment
* Regular use of narcotic pain medication, defined as use on most days of week at any time in the three months prior to surgery
* Significant history of opioid or alcohol abuse or addiction (requiring treatment)
* Delivery of a fetal demise

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Change in postpartum pain control following repair of a second, third, or fourth degree obstetric laceration | Pain control will be assessed at 1, 3, and 7 days after delivery
  The primary goal of the study is to assess how effective the study medication is in providing adequate pain control following repair of a second, third, or fourth degree laceration; therefore, the subjects' post-partum pain will be assessed at various intervals following the repair. On post-partum day one, subjects will be asked questions regarding their pain level in the vaginal area according to the Defense and Veterans Pain Rating Scale, which is an 11-point visual analog pain scale.

SECONDARY OUTCOMES:
Effect on pain medication consumption | Pain medication consumption will be assessed at 1, 3, and 7 days after delivery
  Assess whether the study medication decreases the need for pain medication, specifically opioids, during the post-partum period
Impact pain has on quality of life | Quality of life will be assessed at 1, 3, abd 7 days after delivery
  Evaluate the impact pain has on quality of life comparing the Exparel® and bupivacaine group. Quality of life impact will be evaluated by visual analog supplemental question scale.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Strauchon, DO, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] 2. The Joint Commission. Facts about pain management. Available from: http://www.jointcommission.org/pain_management/. Accessed February 1, 2014.
- [Background] 3. Food and Drug Administration. FDA Drug Safety Communication: Prescription Acetaminophen Products to be Limited to 325 mg Per Dosage Unit; Boxed Warning Will Highlight Potential for Severe Liver Failure. Available from: http://www.fda.gov/drugs/drugsafety/ucm239821.htm. Accessed February 1, 2014.
- [Background] Lyu H, Wick EC, Housman M, Freischlag JA, Makary MA. Patient satisfaction as a possible indicator of quality surgical care. JAMA Surg. 2013 Apr;148(4):362-7. doi: 10.1001/2013.jamasurg.270. PMID 23715968
- [Background] Wheeler M, Oderda GM, Ashburn MA, Lipman AG. Adverse events associated with postoperative opioid analgesia: a systematic review. J Pain. 2002 Jun;3(3):159-80. doi: 10.1054/jpai.2002.123652. No abstract available. PMID 14622770
- [Background] Bramlett K, Onel E, Viscusi ER, Jones K. A randomized, double-blind, dose-ranging study comparing wound infiltration of DepoFoam bupivacaine, an extended-release liposomal bupivacaine, to bupivacaine HCl for postsurgical analgesia in total knee arthroplasty. Knee. 2012 Oct;19(5):530-6. doi: 10.1016/j.knee.2011.12.004. Epub 2012 Jan 28. PMID 22285545
- [Background] Dasta J, Ramamoorthy S, Patou G, Sinatra R. Bupivacaine liposome injectable suspension compared with bupivacaine HCl for the reduction of opioid burden in the postsurgical setting. Curr Med Res Opin. 2012 Oct;28(10):1609-15. doi: 10.1185/03007995.2012.721760. Epub 2012 Sep 3. PMID 22900785
- [Background] Marcet JE, Nfonsam VN, Larach S. An extended paIn relief trial utilizing the infiltration of a long-acting Multivesicular liPosome foRmulation Of bupiVacaine, EXPAREL (IMPROVE): a Phase IV health economic trial in adult patients undergoing ileostomy reversal. J Pain Res. 2013 Jul 18;6:549-55. doi: 10.2147/JPR.S46467. Print 2013. PMID 23901290
- [Background] Vogel JD. Liposome bupivacaine (EXPAREL(R)) for extended pain relief in patients undergoing ileostomy reversal at a single institution with a fast-track discharge protocol: an IMPROVE Phase IV health economics trial. J Pain Res. 2013 Jul 29;6:605-10. doi: 10.2147/JPR.S46950. Print 2013. PMID 23935387
- [Background] Hu D, Onel E, Singla N, Kramer WG, Hadzic A. Pharmacokinetic profile of liposome bupivacaine injection following a single administration at the surgical site. Clin Drug Investig. 2013 Feb;33(2):109-15. doi: 10.1007/s40261-012-0043-z. PMID 23229686
- [Background] Gorfine SR, Onel E, Patou G, Krivokapic ZV. Bupivacaine extended-release liposome injection for prolonged postsurgical analgesia in patients undergoing hemorrhoidectomy: a multicenter, randomized, double-blind, placebo-controlled trial. Dis Colon Rectum. 2011 Dec;54(12):1552-9. doi: 10.1097/DCR.0b013e318232d4c1. PMID 22067185
- [Background] Bergese SD, Ramamoorthy S, Patou G, Bramlett K, Gorfine SR, Candiotti KA. Efficacy profile of liposome bupivacaine, a novel formulation of bupivacaine for postsurgical analgesia. J Pain Res. 2012;5:107-16. doi: 10.2147/JPR.S30861. Epub 2012 May 1. PMID 22570563
- [Background] Chang ZM, Heaman MI. Epidural analgesia during labor and delivery: effects on the initiation and continuation of effective breastfeeding. J Hum Lact. 2005 Aug;21(3):305-14; quiz 315-9, 326. doi: 10.1177/0890334405277604. PMID 16113019
- [Background] Baxter R, Bramlett K, Onel E, Daniels S. Impact of local administration of liposome bupivacaine for postsurgical analgesia on wound healing: a review of data from ten prospective, controlled clinical studies. Clin Ther. 2013 Mar;35(3):312-320.e5. doi: 10.1016/j.clinthera.2013.02.005. Epub 2013 Mar 1. PMID 23453403